CLINICAL TRIAL: NCT01312532
Title: Study of Prosthesis in Total Knee Arthroplasty
Brief Title: Comparing Fixed-bearing Versus Mobile-bearing Prosthesis in Total Knee Arthroplasty: A Prospective Randomized Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Dr. Alireza Yousefy, Associate Professor of Medical Education, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASD-1213-17
Record Dates: First submitted 2011-03-09; First posted 2011-03-10 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2004-06

CONDITIONS: Osteoarthritis
Keywords: Total knee arthroplasty; Fixed-bearing; Mobile-bearing
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fixed-bearing (Other): fixed-bearing device is a kind of prosthesis
  Interventions: Device: fixed-bearing (P.F.C.® Sigma)
- mobile-bearing (Other): mobile-bearing device is a kind of prosthesis
  Interventions: Device: mobile-bearing (P.F.C.® Sigma)

INTERVENTIONS:
Device: fixed-bearing (P.F.C.® Sigma) — P.F.C.® Sigma, DePuy, Johnson & Johnson, Leeds, UK
  Arms: fixed-bearing
Device: mobile-bearing (P.F.C.® Sigma) — P.F.C.® Sigma, DePuy, Johnson & Johnson, Leeds, UK
  Arms: mobile-bearing

SUMMARY:
The purpose of this study is to determine which prosthesis is better in total knee arthroplasty

DETAILED DESCRIPTION:
Theoretical advantages of mobile-bearing devices led surgeons to use these prostheses instead of fixed-bearing devices as traditional implants. This study was designed to compare Fixed-bearing versus Mobile-bearing Prosthesis in Total Knee Arthroplasty through a five-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with expected primary total knee arthroplasty

Exclusion Criteria:

* Mediolateral instability
* Infective arthritis
* Severe deformity
* Revision

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Knee Society Scoring | five years after surgery
  was used for evaluating the function of the knee and high scores indicated better knee function

SECONDARY OUTCOMES:
Pain | five years after surgery
  Pain was evaluated with a Visual Analogue Scale (VAS) with scores ranging from zero to 10ten (0 for no pain and 10 for intolerable pain).

CONTACTS AND LOCATIONS:
Overall Officials: mohammad dehghani, A.Professor, Study Chair — Isfahan University of Medical Sciences
Locations (1):
- Al-zahra university hospital, Isfahan, Isfahan, Iran

REFERENCES:
- See also: Isfahan university of medical sciences — http://mui.ac.ir